CLINICAL TRIAL: NCT05397678
Title: Randomized Trial Evaluating the Non-specific Effects of BCG-Bulgaria and BCG-Denmark in Guinea-Bissau: Effects on Mortality, Morbidity, and BCG Skin Reactions
Brief Title: Trial to Compare BCG-Bulgaria and BCG-Denmark
Acronym: BCGSTRAIN IV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCGSTRAIN IV
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Death; Neonatal; Death, Infant; Morbidity;Newborn; Morbidity;Infant; Non-specific Effects of Vaccines
Keywords: Bacillus Calmette-Guérin; BCG vaccine; Non-specific effects of BCG; Heterologous effects; Maternal immune priming; Maternal BCG scar
MeSH Terms: conditions — Perinatal Death; Infant Death

STUDY DESIGN:
Intervention Model Description: Outcome assessor-blinded RCT
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Following informed consent, the child's mother/guardian selects, from a stack of envelopes, a closed envelope that contains a sealed randomization lot indicating allocation to either BCG-Denmark or BCG-Bulgaria. The mother, inclusion assistant and vaccinator will thus not be blinded to the intervention allocation. All assistants assessing outcomes during follow-up procedures and providers of care will be blinded to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG-Denmark (Experimental): Infants randomized to receive BCG-Denmark at discharge from the Maternity Ward will receive one 0.05 ml infant dose of Mycobacterium bovis BCG live-attenuated BCG-AJ vaccine by intradermal injection in the left deltoid region. Dependent on national supply, oral polio vaccine will be co-administered.
  Interventions: Biological: BCG-Denmark
- BCG-Bulgaria (Active Comparator): Infants randomized to receive BCG-Bulgaria at discharge from the Maternity Ward will receive one 0.05 ml infant dose of Mycobacterium bovis BCG live-attenuated BCG-Bulgaria vaccine by intradermal injection in the left deltoid region. Dependent on national supply, oral polio vaccine will be co-administered.
  Interventions: Biological: BCG-Bulgaria

INTERVENTIONS:
Biological: BCG-Denmark — AJ vaccines, Copenhagen 1331 strain
  Other Names: BCG-AJ; BCG-SSI
  Arms: BCG-Denmark
Biological: BCG-Bulgaria — BB-NCIPD Ltd., BCG-SL 222 Sofia strain
  Other Names: BCG-Sofia
  Arms: BCG-Bulgaria

SUMMARY:
The trial will be a two-year outcome assessor-blinded RCT at the maternity ward of Hospital Simão Mendes (HNSM) in urban Bissau, Guinea-Bissau to compare vaccination with Bacillus Calmette-Guérin (BCG) Danish strain (AJ Vaccines, Copenhagen 1331 strain) versus BCG-Bulgaria (BB-NCIPD, BCG-SL 222 Sofia strain) 1:1 in 15,000 infants with respect to mortality, morbidity and case-fatality rate during hospital admission. The trial will also examine the association between BCG strains and BCG skin reaction kinetics and characteristics.

As a secondary aim, this large study will be used to further evaluate the role of maternal BCG immune priming for overall health, since there are indications that the maternal BCG scar status influences offspring health outcomes.

DETAILED DESCRIPTION:
This two-year outcome assessor-blinded RCT will be conducted at the maternity ward of hospital Simão Mendes (HNSM) in urban Bissau, Guinea-Bissau to compare BCG-Denmark versus BCG-Bulgaria 1:1 in 15,000 infants with respect to mortality, morbidity and case-fatality rate during hospital admission.

The trial will also examine the association between BCG strains and BCG skin reaction kinetics and characteristics.

HYPOTHESES

The investigators aim to investigate the following hypotheses:

1. Compared with BCG-Bulgaria, receiving BCG-Denmark is associated with

   1. a 35% reduction in all-cause deaths and
   2. a 50% lower case-fatality rate for hospitalized infants.
2. BCG-vaccinated infants have lower mortality and in-hospital case-fatality risk if the mother has a BCG scar than if the mother does not have a BCG scar.
3. BCG-Denmark is associated with more favorable early-life BCG skin reaction kinetics (prevalence, type, size)

METHODS Setting: The RCT will be carried out by the BHP in close collaboration with the Maternity Ward of HNSM in Bissau. A dedicated BHP team registers births and oversees all vaccinations at the Ward, where BHP has conducted a series of RCTs since 2002, with the aim of improving early-life health outcomes. The BHP maintains a Health and Demographic Surveillance System (HDSS) comprising approx. 100,000 individuals in the capital Bissau.

Inclusion: Neonates born at the HNSM Maternity Ward and neonates referred to the ward for vaccination from the adjacent Pediatric Ward, the Neonatal Intensive Care Ward and the Maternity Center receive their neonatal vaccines at the Maternity Ward and are eligible for participation in the study. Mothers/guardians to infants eligible for the study will receive an oral study explanation in Portuguese Creole and a written explanation in Portuguese. Provided that oral consent is obtained, the mother/guardian signs a written consent form; if the mother or guardian is illiterate, a fingerprint can be provided to confirm participation. The family can request that their child leaves the trial at any time. Infants that are not eligible for participation or whose mother/guardian declines participation will be registered and provided the routine vaccinations by the study team (standard practice). Information on maternal and paternal BCG scar status, scar size, mid-upper-arm circumference and socioeconomic factors will be collected during the inclusion procedure.

Telephone contact information for the mother, the father and family members and/or persons living in the same house are recorded at inclusion. Infants for whom only 0 or 1 telephone numbers are available at inclusion will be transported home by a BHP car, when possible, to secure more telephone numbers, provided consent has been obtained and the family lives in greater Bissau. Similarly, infants from the HDSS with incomplete address information will be transported home, when possible, to correctly register the address of the family house. BCG will be provided at discharge for all infants at the ward and a sticker is placed on the vaccination card of all neonates assessed for eligibility to the study, regardless of participation. This sticker provides access to free consultations at three health centers located in the HDSS with essential drugs provided free of charge.

Randomization: Following informed consent, the mother selects, from a stack of envelopes, a closed envelope that contains a sealed randomization lot indicating allocation to either BCG-Denmark or BCG-Bulgaria. The mother, inclusion assistant and vaccinator will thus not be blinded to the intervention allocation. The envelope and randomization lot are opened, and the lot is stapled to the inclusion form. Randomization lot envelopes are prepared by a senior staff supervisor in separate bundles of 40 for each sex.

Vaccination: The infant is vaccinated intradermally with 0.05 ml of the allocated BCG strain in the left upper deltoid, followed by vaccination with OPV. OPV is provided via the National Vaccination Program; if OPV is in shortage, only BCG vaccination will be provided.

Follow-up: All assistants assessing outcomes during the follow-up procedures outlined below will be blinded to the randomization allocation.

Follow-up takes place through three mechanisms:

A) All enrolled infants with a telephone number recorded at inclusion: Family telephone interview at one week, six weeks and six months of age.

Families are telephoned to register dates and outcomes of hospital admissions and whether the child is alive. If the child died, the mother/guardian is briefly asked about symptoms and whether the death occurred at home or at a hospital. Information on adherence to the six-week vaccination schedule, infant BCG skin reaction status (yes/no, type of skin reaction) and adverse events is also collected. Priority will be given to interview the mother or father of the child when possible. Based on previous experiences summarized in Table 5, 99% of families provided at least one telephone number at inclusion and the overall follow-up rate by telephone is approx. 95%.

B) Cohort of BHP HDSS infants: home visit during the first two months of life. With the proposed sample size of 15,000 infants and an estimated 15% residing in the HDSS study area, the study will include approximately 2,250 children from the HDSS. In addition to follow-up within the routine surveillance system maintained by the investigators, these children will receive one additional home visit between one week and eight weeks of age. At the visit, trial assistants will collect data on mortality, morbidity, BCG skin reaction status, type and size, adverse events and maternal and paternal BCG scar status and size (if not collected at inclusion). The visit is conducted between one and eight weeks of age to collect data regarding the kinetics of early BCG skin reactions (prevalence, type).

C) All enrolled infants: Registration of admissions and consultations at the HNSM pediatric ward.

Admissions, diagnoses and outcomes at the pediatric ward are documented by a BHP team on all days of the year. Parental names and telephone numbers are registered for all admissions. For approximately 60% of infant admissions, data from the child's health card is documented during the admission, ensuring registration of the child's unique study ID for later data linkage. To identify the remaining admissions not registered with the unique study ID, a previously validated standardized systematic database linkage and search algorithm will be applied.

Sample size:

There are approx. 7,000 childbirths per year at the maternity ward of the HNSM and an additional 500-600 neonates not born at HNSM are vaccinated there each year. With an expected monthly inclusion rate of 600 infants based on previous experiences, the investigators expect to be able to include at least 15,000 children, i.e. 7,500 in each BCG strain group, during an expected timeframe of approx. two years for inclusion procedures and an additional six months for follow-up procedures.

Analyses:

The mortality and morbidity data will be analyzed as intention-to-treat in Cox regression models with age as the underlying time variable, i.e. with complete adjustment for age. In-hospital case-fatality rates between BCG strains will be compared using binomial regression. In case an OPV or other campaigns with potential immune stimulatory effects occurs during the study period, the main comparison of the two strains and of the effects of maternal BCG scarring on infant outcomes will be conducted by censoring all children on the first day of the campaign, to exclude any interaction of the campaign with the BCG strains.

As sensitivity analyses, an analysis where events occurring on the day of BCG vaccination are omitted will be conducted. An analysis of main outcomes excluding neonates that were admitted at the pediatric or NICU ward before inclusion will also be conducted. In case there are shortages of OPV and thus neonates included that do not receive OPV-0, an analysis of main outcomes by receipt of OPV-0 will be conducted.

The investigators will conduct explorative analyses evaluating effects of the BCG strains by post-vaccination wheal size (<5mm vs >5mm), sex, and vaccinator.

All analyses will be conducted overall and stratified by maternal BCG scar status and sex. The investigators will conduct an analysis of the independent effect of the maternal scar status on trial outcomes with adjustment for possible associations between socioeconomic factors and maternal BCG scarring that can also affect the mortality risk in the offspring.

Trial vaccines:

In the event that BCG-Denmark and/or BCG-Bulgaria is available via the Nationwide Program of Vaccination (EPI) in Guinea-Bissau and thus provided to the BHP team at HNSM, these vaccines will be considered equivalent and used as trial vaccines. If not available, the BCG vaccines will be acquired from AJ Vaccines (BCG-Denmark, Copenhagen 1331 strain) and BB-NCIPD (BCG-Bulgaria, BCG-SL 222 Sofia strain). If there are unforeseen difficulties procuring the trial vaccines, BCG-Bulgaria can be substituted with either of the following genetically similar strains: BCG-Russia (Russian BCG-I strain, Microgen, Russia) or BCG-Russia (Serum Institute of India, Pune, India). BCG-Denmark can be substituted with either of the following: BCG-GreenSignal (Copenhagen 1331, GreenSignal Bio Pharma), BCG-Chennai (Copenhagen 1331, BCG Vaccine Laboratory Chennai), or BCG-Tokyo (Tokyo 172-1 strain, Japan BCG laboratory).

Ethical considerations:

The proposed study will randomize children to two BCG strains that are prequalified and distributed by UNICEF and used in both Guinea-Bissau and the rest of the world. Previous studies from the investigators have shown that providing BCG vaccination at discharge is safe and beneficial. Oral and written informed consent will be obtained in all cases. The BHP offers medical consultations at two HDSS health centers to all infants assessed for eligibility, independent of eligibility or whether the mother/guardian chose to participate or not. Essential medications are available through the PIMI program free-of-charge, but in case they run out or the PIMI program is discontinued during the trial, BHP offers essential drugs as a back-up. The mothers are encouraged to bring their child for consultation at a health center if their child develops lymphadenitis.

The study protocol will be submitted for approval by the Ethical Committee in Guinea-Bissau and to the Central Ethical Committee in Denmark for consultative approval. A local clinical monitor will be appointed to oversee the study.

ELIGIBILITY:
Inclusion criteria:

- Healthy infants under one year of age who are vaccinated at the HNSM maternity ward.

Exclusion criteria:

* Infants who have already received either BCG or oral polio vaccine (OPV)
* Infants who are moribund due to gross malformation or acute illness (about to die or be transferred to the pediatric ward according to the local health physician assessment); the latter children can be recruited when they are discharged from the pediatric ward or the neonatal intensive care unit.

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15000 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality risk | Six weeks of age
  Deaths from all-causes

SECONDARY OUTCOMES:
All-cause mortality risk | One week of age
  Deaths from all-causes
All-cause mortality risk | Six months of age
  Deaths from all-causes
In-hospital case-fatality rate | Six weeks of age
  Deaths occurring among infants admitted at the Hospital Nacional Simão Mendes pediatric ward
In-hospital case-fatality rate | Six months of age
  Deaths occurring among infants admitted at the Hospital Nacional Simão Mendes pediatric ward
Hospital admission from all causes | Six weeks of age
  Admissions at the Hospital Nacional Simão Mendes pediatric ward
Hospital admission from all causes | Six months of age
  Admissions at the Hospital Nacional Simão Mendes pediatric ward
BCG skin reaction prevalence and type | Assessed at one week of age
  All enrolled infants reached by telephone follow-up.
BCG skin reaction prevalence and type | Assessed at six weeks of age
  All enrolled infants reached by telephone follow-up.
BCG skin reaction prevalence and type | Assessed at six months of age
  All enrolled infants reached by telephone follow-up.
BCG skin reaction prevalence, type and size | Assessed at one home visit per child conducted during the first eight weeks of life
  Subgroup of infants residing within the BHP Health and Demographic Surveillance System

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Professor, Principal Investigator — Bandim Health Project; Christine Stabell Benn, Professor, Study Chair — University of Southern Denmark and Bandim Health Project; Frederik Schaltz-Buchholzer, MD, PhD, Study Director — University of Southern Denmark and Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data with a data dictionary can be shared after approval of a data-sharing proposal sent to Professor Christine Stabell Benn (cbenn@health.sdu.dk).